CLINICAL TRIAL: NCT00582621
Title: Ascertainment of Families for Genetic Studies of Familial Lymphoproliferative Disorders
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Montefiore Medical Center (Other); St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 00-069
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Leukemia; Multiple Myeloma; Colon Cancer; Renal Cancer
Keywords: Genetic Studies; 00-069; blood; saliva; buccal cell
MeSH Terms: conditions — Lymphoma; Leukemia; Multiple Myeloma; Colonic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or alternatively, subjects may provide a saliva or buccal cell sample

SUMMARY:
The purpose of this study is to better understand the genetic causes of Hodgkin's disease (a kind of lymphoma) and non-Hodgkin's lymphoma, as well as multiple myeloma, leukemia, and related diseases. The doctors have identified the patient because 1) they have had a lymphoproliferative disorder such as lymphoma, leukemia, or multiple myeloma, and have a family member with one of these disorders or 2) they are a member of a family with a lymphoproliferative disorder, including Hodgkin's disease and/or, non-Hodgkin's lymphoma or a second cancer after Hodgkin's disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a personal and/or family history of lymphoma or lymphoproliferative disease B-cell malignancies, or multiple myeloma referred for study participation, or MSK patients referred from to the MSKCC outpatient clinics of the Lymphoma, Multiple Myeloma, or Leukemia Services in the Department of Medicine in consultation for treatment who are found on routine history or through a Family History Questionnaire (FHQ) (Appendix A). Individuals who have relatives or members of successive generations of the family affected with Hodgkin's disease, non-Hodgkin's lymphoma, lymphoid leukemia, multiple myeloma other lymphoproliferative disease prostate or pancreatic cancers, or other conditions suggesting hereditary cancer at the discretion of the MSKCC Principal Investigator. Patients with lymphoma, associated with colon and renal cancer will be eligible for DNA storage through this protocol. Family members or probands with Hodgkin's disease who are women who received therapeutic irradiation for Hodgkin's disease" or who developed secondary cancers after Hodgkin's disease are also eligible for participation.
* The criteria for eligibility are broad because the ascertainment by the computerized FHQ does not allow for resolution of different types of lymphoma or different types of leukemia. Patient recall of this information is also imprecise. More accurate family history information will be obtained upon contact of family members and diagnoses will be verified by obtaining pathologic documentation. The spectrum of familial lymphoproliferative syndromes (LPS) may include all types of lymphoma as well as chronic lymphocytic leukemia. This is an additional reason to have a broad eligibility. Subset analysis will be performed on specific types of lymphoid neoplasms. DNA of patients with a family history of lymphoma who have consented to protocol 93-102 ("Ascertainment of Peripheral Blood or Saliva Samples for Genetic Epidemiology Studies of Familial Cancers") will also be eligible for inclusion in this study.
* Family members of probands including patients, sisters, brothers, halfbrothers and sisters, sons, daughters, grandparents, as well as aunts and uncles are also eligible. An effort will be made to ascertain all living affected and unaffected living relatives in the affected lineage. An emphasis will be on affected sibling pairs and both parents, if alive.
* As this study involves research that presents no greater than minimal risk to children (see Sec. 46.404 of Federal Regulations part 46), minors are also eligible for participation. The assent of any minor should be obtained before the patient is enrolled into this study, as well as the consent of the legal guardian.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinical Genetics Service at MSKCC or to the MSKCC outpatient clinics of the Lymphoma, Multiple Myeloma or Leukemia Services in the Department of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2000-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To establish a collection of DNA and frozen lymphocytes for the purpose of facilitating genetic laboratory investigations of familial lymphoid neoplasms. | 2 years

SECONDARY OUTCOMES:
To perform linkage and candidate gene studies on informative families for the purpose of identifying novel lymphoproliferative syndrome (LPS) predisposition genes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org